CLINICAL TRIAL: NCT03915080
Title: Optimizing the Use of Prophylaxis in Patients With Severe Haemophilia A Using PK Measurement (myPKFiT)
Brief Title: Optimizing the Use of Prophylaxis in Patients With Severe Haemophilia A
Acronym: myPKFiT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20160920
Record Dates: First submitted 2016-12-13; First posted 2019-04-16 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oktokog alpha (Advate) (Other): Personalized treatment according to individual PK using intravenous injection of oktokog alpha with dose and dose interval according to MyPKFIT and phenotypic evaluation.
  Interventions: Drug: Oktokog alpha

INTERVENTIONS:
Drug: Oktokog alpha — adjusting dose and dose interval according to MyPKFIT

SUMMARY:
MyPKFiT is a web-based application recently developed by Baxalta for the use in patients treated with Advate. MyPkFit has its basis in Bayesian forecasting, which allows estimation of individual PK parameters by a sparse sampling schedule, where only 2-3 samples are taken between 4 and 48 hours post infusion. With myPKFiT, it will, therefore, be possible to define an individual PK curve for each patient based on just a few sampling points and hence, taking the bleeding phenotype and the life style into account, potentially adjust the prophylactic treatment accordingly to optimize cost-effectiveness.

DETAILED DESCRIPTION:
As detailed in brief summary patients will, after accurate information verbally and written according to ethics approval, report bleeding events during previous 6 months. Blood samples are taken, FVIII analyzed (Advate patients) and the individual PK curve determined using MyPKFit. The curve will be discussed together with the patient and levels related to bleed events determined. If needed dose adjustment is done based on the curve. After a further 6 month follow-up bleeds will again be evaluated as well as factor consumption. In this way a better personalized treatment based on PK and clinical phenotype will hopefully be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with severe hemophilia A (FVIII:C <1 %), being treated with Advate for more than 50 exposure days (EDs

Exclusion Criteria:

* Current evidence of inhibitor as measured by the Nijmegen-modified Bethesda assay
* Use of another investigational FVIII product in the previous month

Ages: 1 Year to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-12; Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
PK measurement to individualize replacement therapy | 3 years
  To evaluate whether PK measurement by myPKFiT and the calculation of an individualized PK profile may allow the treating physician to personalize and optimize the treatment of patients with haemophilia A to minimize the number of bleeds in a cost-effective way without diminishing compliance.
PK measurement to influence FVIII consumption | 3 years
  2. To calculate whether optimization of treatment by use of MyPKFiT, as described in primary objective 1, result in change of total FVIII consumption and extra doses given before and after visit 1. Measurements are T1/2, area under the curve
Specific pharmacokinetic parameters to analyze | 3 years
  Biological half-life of infused FVIII product will be measured in hours. Area under the curve (AUC)will be given in IUxh/dL

SECONDARY OUTCOMES:
Signs of hemophilic arthropathy | 3 years
  1. To identify and characterize and sign of arthropathy by ultrasound sound evaluation of the synovium, cartilage and bone according to the HEAD-US score of ankle, knee and elbows visit 1 and 2 and correlate this to the treatment provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö Centre for Thrombosis and Haemostasis, Malmo, Sweden